CLINICAL TRIAL: NCT03580083
Title: A Phase I/II Multicenter, Open-Label Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of Intracisternal RGX-111 in Subjects With Mucopolysaccharidosis Type I
Brief Title: RGX-111 Gene Therapy in Patients With MPS I
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: REGENXBIO Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGX-111-002
Record Dates: First submitted 2018-06-18; First posted 2018-07-09 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Mucopolysaccharidosis Type I (MPS I); Hurler Syndrome; Hurler-Scheie Syndrome
Keywords: MPS I , gene therapy, Hurler, Hurler- Scheie
MeSH Terms: conditions — Mucopolysaccharidosis I

STUDY DESIGN:
Intervention Model Description: Sequential Assignment Dose escalation
Masking Description: Open-Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose 1; 1x10^10 GC/g brain mass of RGX-111 (Experimental)
  Interventions: Genetic: RGX-111
- Dose 2; 5x10^10 GC/g brain mass of RGX-111 (Experimental)
  Interventions: Genetic: RGX-111

INTERVENTIONS:
Genetic: RGX-111 — Recombinant adeno-associated virus serotype 9 capsid containing α-L-iduronidase expression cassette

SUMMARY:
RGX-111 is a gene therapy which is intended to deliver a functional copy of the α-L-iduronidase (IDUA) gene to the central nervous system. This is a safety and dose ranging study to determine whether RGX-111 is safe and tolerated by patients with MPS I.

DETAILED DESCRIPTION:
Mucopolysaccharidosis type I (MPS I) is a rare recessive genetic disease caused by a deficiency of α-L-iduronidase (IDUA) leading to an accumulation of glycosaminoglycans (GAGs) in tissues of patients with MPS I. While currently available therapies, enzyme replacement therapy (ERT) and hematopoietic stem cell transplantation (HSCT), provide clinical benefit over untreated disease progression, they still possess significant limitations. ERT does not cross the blood-brain barrier and, therefore, does not treat the central nervous system (CNS) effects of the disease, and HSCT has clinically relevant morbidity and mortality and is not able to completely treat the CNS effects. RGX-111 is designed to deliver a functioning gene enabling the production of IDUA in the brain. This is a Phase I/II, first-in-human, multicenter, open-label, dose escalation study of RGX-111. Up to 11 subjects with MPS I will be treated in 2 dose cohorts and will receive a single dose of RGX-111. Safety will be the primary focus for the initial 24 weeks after treatment (primary study period) whereupon, subjects will continue to be assessed (safety and efficacy) for up to a total of 104 weeks following treatment with RGX-111.

ELIGIBILITY:
Inclusion Criteria:

1. Has documented evidence of CNS involvement due to MPS I or documented diagnosis of severe MPS I
2. Subjects who have had HSCT may be enrolled in the study if the PI, medical monitor, and sponsor agree that he/she can participate in the study.

Exclusion Criteria:

1. Has contraindications for intracisternal and intracerebroventricular injection or lumbar puncture.
2. Has contraindications for immunosuppressive therapy.
3. Has neurocognitive deficit not attributable to MPS I or diagnosis of a neuropsychiatric condition.
4. Received intrathecal (IT) laronidase at any time and experienced a significant AE considered related to IT administration
5. Has received intravenous (IV) laronidase at any time and experienced a significant AE considered related to IV administration.
6. Received any investigational product within 30 days of Day 1 or 5 half-lives before signing of the Informed Consent Form (ICF), whichever is longer.
7. Has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 × upper limit of normal (ULN) or total bilirubin >1.5 × ULN at screening unless the subject has a previously known history of Gilbert's syndrome and a fractionated bilirubin that shows conjugated bilirubin <35% of total bilirubin.

Min Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Safety: Number of participants with treatment-related adverse events and serious adverse events | 24 Weeks
  Number of participants with treatment-related adverse events and serious adverse events

SECONDARY OUTCOMES:
Safety: Number of participants with treatment-related adverse events | 104 Weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE (Version 4.03)
Change in neurodevelopmental parameters | Baseline, Week 24, Week 52, Week 78, Week 104
  As measured by the Wechsler Abbreviated Scale of Intelligence, 2nd Edition (WASI-II).Based on their mean age equivalence score on the Vineland Adaptive Behavior Scales (#7) the subject will be assessed using the WASI-II ( for scores of >/= 72 months).
Change in neurodevelopmental parameters | Baseline, Week 24, Week 52, Week 78, Week 104
  As measured by the Bayley Scale of Infant and Toddler Development, Third Edition (Bayley-III). Based on their mean age equivalence score on the Vineland Adaptive Behavior Scales (#7) the subject will be assessed using the BSID-III (for scores of </ = 36 months or >36 months to <42 months) .
Change in neurodevelopmental parameters | Baseline, Week 24, Week 52, Week 78, Week 104
  As measured by the Wechsler Preschool and Primary Scales of Intelligence, Fourth Edition (WPPSI-IV). Based on their mean age equivalence score on the Vineland Adaptive Behavior Scales (#7) the subject will be assessed using the WPPSI-IV (for scores >36 months to < 42 months OR for scores of >/= 42 months and <72 months or >36 months to <42 months and unable to complete BSID-III (#4)) .
Change in neurodevelopmental parameters | Baseline, Week 24, Week 52, Week 78, Week 104
  Change from baseline in neurodevelopment parameters of attention as measured by the Tests of Variables of Attention, Version 9 (TOVA) if able to complete the WASI-II (as defined in #3).
Change in adaptive behavior | Baseline, Week 12, Week 24, Week 36, Week 52, Week 78, Week 104
  Change in baseline in adaptive behavior as measured by the Vineland Adaptive Behavior Scales, Third Edition (VABS-III)
Vector shedding | Baseline, Week 1, Week 4, Week 8, Week 16, Week 24
  As measured by vector concentration (quantitative polymerase chain reaction [qPCR] to RGX-111 deoxyribonucleic acid [DNA]) in CSF, serum, and urine

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil
- Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De BP, Rosenberg JB, Selvan N, Wilson I, Yusufzai N, Greco A, Kaminsky SM, Heier LA, Ricart Arbona RJ, Miranda IC, Monette S, Nair A, Khanna R, Crystal RG, Sondhi D. Assessment of Safety and Biodistribution of AAVrh.10hCLN2 Following Intracisternal Administration in Nonhuman Primates for the Treatment of CLN2 Batten Disease. Hum Gene Ther. 2023 Sep;34(17-18):905-916. doi: 10.1089/hum.2023.067. PMID 37624739